CLINICAL TRIAL: NCT02155998
Title: A Non-interventional Study of Postoperative or Post-Radiation trEatment Habits in Locally adVanced Prostate Cancer patiENTs (High Risk)- PREVENT
Brief Title: Non-Interventional Study PREVENT
Acronym: PREVENT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ORU-XXX-2014/2
Record Dates: First submitted 2014-06-03; First posted 2014-06-04 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Postoperative or Postradiation Adjuvant Androgen Deprivation Therapy in Locally Advanced Prostate Cancer (High and Very High Risk) Patients
Keywords: prostate adenocarcinoma, locally advanced prostate cancer with high and very high risk of recurrence, adjuvant endocrine treatment, prostate specific antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PREVENT study patients: Patients with locally advanced prostate cancer with high and very high risk of recurrence, who underwent surgery or radiotherapy within 3 months prior to enrolment, 18 years and older, consented to participate in this non-interventional study, being treated for prostate cancer in the oncology institutions / departments in the Russian Federation.

SUMMARY:
This is a multicentre, non-interventional, prospective study to be carried out in representative medical institutions in order to get the information on administration of postoperative and post-radiation adjuvant androgen deprivation therapy (including "go" / "no go" decision, regimens, dosages and duration) used in locally advanced prostate cancer patients with high and very high risk of recurrence in Russia.

DETAILED DESCRIPTION:
This is a multicentre, non-interventional, prospective study to be carried out in representative medical institutions in order to get the information on administration of postoperative and post-radiation adjuvant androgen deprivation therapy (including "go" / "no go" decision, regimens, dosages and duration) used in locally advanced prostate cancer patients with high and very high risk of recurrence in Russia.

No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

It is planned to enrol 200 subjects in up to 30 sites in Russian Federation. The average number of patients per site is planned as 6 - 10; there are no restrictions on minimum and maximum number of subjects per site in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The voluntarily given informed consent, confirmed by the Informed Consent Form, properly signed by both the subject and the investigator.
2. Locally advanced stage of PCa (stage T3-T4, Nx-N0, M0: prostate adenocarcinoma with extracapsular invasion (T3a) or invasion to the seminal vesicles (T3b), invasion to adjacent structures (T4) but without lymphatic invasion (N0) nor metastasis (M0))
3. Prostatectomy or radiotherapy completed within 3 months prior to the study enrolment
4. High (T3a or Gleason score = 8-10 or PCA >20 ng/ml) and very high (T3b-T4) risk of recurrence
5. Histologically confirmed diagnosis of prostate adenocarcinoma

Exclusion Criteria:

1. Patients participating in clinical trials
2. Any medical condition which on the opinion of the investigator may interfere with the patient's participation in the study, e.g. severe non-malignant concomitant disease which can affect life expectancy
3. Evidence of metastatic disease on imaging studies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients with locally advanced prostate cancer with high and very high risk of recurrence, who underwent surgery or radiotherapy within 3 months prior to enrolment, 18 years and older, consented to participate in this non-interventional study, being treated for prostate cancer in the oncology institutions / departments in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-07-16 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of adjuvant endocrine therapy: drugs used for androgen deprivation therapy, regimen, dose, duration | up to 15 months after LSI
  Evaluation of adjuvant endocrine therapy: drugs used for androgen deprivation therapy, regimen, dose, duration

SECONDARY OUTCOMES:
Data collection of patients characteristics (age, race, co-morbidities, family history of prostate cancer) | up to 15 months after LSI
  Data collection of patients characteristics (age, race, co-morbidities, family history of prostate cancer)
Data collection of disease information ( disease stage - TNM, histology, Gleason score, PSA level, prior prostate cancer surgery/radiotherapy -types, imaging techniques, neoadjuvant and adjuvant therapy(medications by groups, orchidectomy) | up to 15 months after LSI
  Data collection of disease information ( disease stage - TNM, histology, Gleason score, PSA level, prior prostate cancer surgery/radiotherapy -types, imaging techniques, neoadjuvant and adjuvant therapy(medications by groups, orchidectomy)
Proportion of patients with double increase in PSA level during 1 year follow-up | up to 15 months after LSI
  Proportion of patients with double increase in PSA level during 1 year follow-up
Proportion of progression-free patients after 1 year follow-up | up to 15 months after LSI
  Proportion of progression-free patients after 1 year follow-up
Proportion of patients with disease progression after 1 year follow-up | up to 15 months after LSI
  Proportion of patients with disease progression after 1 year follow-up
Proportion of patients having biochemical relapse after 1 year follow-up | up to 15 months after LSI
  Proportion of patients having biochemical relapse after 1 year follow-up
Proportion of patients having clinical relapse (local or metastatic) after 1 year follow-up | up to 15 months after LSI
  Proportion of patients having clinical relapse (local or metastatic) after 1 year follow-up
Evaluation of deaths among BRCAm+ patient | up to 15 months after LSI
  Evaluation of deaths among BRCAm+ patient

CONTACTS AND LOCATIONS:
Overall Officials: Karin Otter, Study Director — AstraZeneca; Boris Alexeev, Principal Investigator — Moscow Research Institute of Oncology named after PA Herzen; Vsevolod Matveev, Principal Investigator — Russian Cancer Research Center named after NN Blokhin
Locations (14):
- Russia (14):
  - Research Site, Balashikha
  - Research Site, Belgorod
  - Research Site, Izhevsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Tula
  - Research Site, Tyumen
  - Research Site, Vladimir

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3020&filename=PREVENT_%20NIS%20PrimaryReport_Final_20%2003%202019_with%20masked%20information.pdf